CLINICAL TRIAL: NCT01312623
Title: Organ Protection by Remote Ischemic Preconditioning for Surgical Treatment of Pediatric Congenital Heart Disease
Acronym: RIPHeart
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated, because it is not possible to recruit enough participants
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Axel Fudickar, Dr. med., University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudickar5
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Heart Ischemia; Cerebral Ischemia
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote ischemic preconditioning (Experimental): Remote ischemic preconditioning at the left leg.
  Interventions: Other: Remote ischemic preconditioning
- Control (No Intervention): No ischemic preconditioning

INTERVENTIONS:
Other: Remote ischemic preconditioning — Remote ischemic preconditioning at the left leg.
  Arms: Remote ischemic preconditioning

SUMMARY:
Cardiac surgery is associated with risk of perioperative inflammation and ischemia leading to cerebral and myocardial morbidity and mortality. Ischemic preconditioning by repetitive ischemic episodes at an organ can reduce damage resulting from consecutive prolonged ischemia in that organ. Remote ischemic preconditioning is defined as ischemic preconditioning by repetitive ischemic episodes of an organ remote from the organ to be protected, e.g. ischemic episodes of a limb can reduce ischemic damage of the heart. Animal studies as well as human studies have shown that ischemic preconditioning can protect the heart from intraoperative ischemia. Remote preconditioning by repetitive limb ischemia has been applied in humans in some studies.12-14 However, the published data is not yet sufficient to support evidence based recommendations for clinical practice. In particular, available data regarding the influence of remote preconditioning on inflammatory and ischemic damage of brain and heart in children following surgery of congenital heart disease are limited. Hence, this prospective, controlled and randomized study was designed to perform remote ischemic preconditioning in children after induction of anesthesia for pediatric heart surgery and to investigate the effect on postoperative organ function in comparison to a control group.

DETAILED DESCRIPTION:
Arterial blood flow to the right leg of the patients is interrupted by inflating a cuff around the thigh up to a pressure of 15 mmHg above the systolic blood pressure for five minutes. Thereafter the pressure is released for another five minutes and the procedure is repeated fourfold. Cerebral and myocardial damage are examined by postoperative laboratory exams in comparison to preoperative baseline values. In addition to this, systemic immune response, renal function, duration of intensive care and time to discharge from hospital are compared between groups. Mechanisms of remote preconditioning are investigated by analyzing gene expression in human heart tissue obtained during surgery and in leukocytes.

The investigation is not associated with any known risks for the children.

ELIGIBILITY:
Inclusion Criteria:

* congenital heart surgery

Exclusion Criteria:

* hypoplastic left heart syndrome

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
serum troponin T | 48 hours
  Serum troponin T is measured 8, 16 and 24 hours after end of surgery. Values of serum troponin T are compared between remote ischemic preconditioning group and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Fudickar, Dr., Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No